CLINICAL TRIAL: NCT06627725
Title: The Effect of Patient-Family Communication Via Audio Recording on Anxiety, Depression, and Satisfaction of Cardiovascular Intensive Care Unit (CICU) Patients&Amp;Amp;Amp;#39; Relatives: Randomized Controlled Trial
Brief Title: The Effect of Patient-Family Communication Via Audio Recording
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Kalkan Uğurlu (Other)
Responsible Party: Sponsor-Investigator, Yasemin Kalkan Uğurlu, Assit Prof., Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1988
Record Dates: First submitted 2024-09-28; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Anxiety Depression (Mild or Not Persistent); Satisfaction With Care
Keywords: Anxiety; Family; Depression; Satisfaction; intensive care unit
MeSH Terms: conditions — Anxiety Disorders; Lymphoma, Follicular; Depression; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Interventional Study Model.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The voice message prepared by a patient's relative, decided by the patient's family members, was recorded using a voice recorder. Before the voice message was recorded, the researcher met with the patient's relative and gave preliminary information about the message content (Table 1) in order to prevent the message from negatively affecting the patient. In the study, care was taken to ensure that the messages to be played to the patient were between 3-5 minutes and simple terms that could be understood by individuals with low educational level were used. The patient's relatives recorded the messages they wanted to convey to the patient with a voice recorder. The voice message was played to the patient by the researcher using a music pillow in the CICU . After the condition of the patient in the intervention group stabilized, a pretest (IIF, HADS, VAS-A, FS-ICU) was administered to the patient's relative, then a voice recording was prepared and the patient's relative's voice recording
  Interventions: Behavioral: Patient-Family Communication
- Control (No Intervention): After the condition of the patients in the control group stabilized, a pretest (IIF, HADS, VAS-A, FS-ICU) was administered to the relatives. Afterwards, the relatives were routinely informed about the patient's general condition, treatment process, and needs.

INTERVENTIONS:
Behavioral: Patient-Family Communication — Patient-Family Communication
  Arms: intervention

SUMMARY:
The study was conducted as a randomized controlled blinded study. The sample consisted of 55 patient relatives (27 in the experimental group and 28 in the control group). The patient's relatives in the experimental group said what they wanted to say to their patient in line with the content determined by the researchers and recorded it using a voice recorder. The researcher played the recorded message to the patient, and the patient's feedback was conveyed to the patient's relative.

DETAILED DESCRIPTION:
Visitor restrictions in coronary intensive care units (CICUs), which make it difficult for relatives to communicate with and support their patients, can lead to negative emotional reactions such as anxiety, depression and anger in family members. This study was conducted to determine the effect of playing the voice recording of the relatives to the patients hospitalized in CICU on the anxiety, depression and satisfaction levels of the relativesThe study was conducted as a randomized controlled single blinded study. The sample consisted of 55 patient relatives (27 in the experimental group and 28 in the control group). The patient's relative in the experimental group said what they wanted to say to their patient in line with the content determined by the researchers and recorded it using a voice recorder. The recorded message was played to the patient by the researcher and the feedback of the patient was conveyed to the patient's relative by the researcher. The relatives of the patients in the control group were routinely informed. The "Patient Relative Introduction Form", "Hospital Anxiety Depression Scale (HADS)", "Visual Analog Scale-Anxiety (VAS-A)" and "Satisfaction Scale of Families of Patients Hospitalized in Intensive Care Unit (FS-ICU)" were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Turkish,
* Being a first-degree relative of a patient hospitalized in the CICU with AMI.

Exclusion Criteria:

* Hearing and speech problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
The Hospital Anxiety Depression Scale | 10 minutes
  The scale consists of 14 items, seven items measure anxiety (HAD-A) and the other seven items measure depression (HAD-D). The scale is a four-point Likert-type scale with a total scoe of 0-42.
Visual Analog Scale | 2 minutes
  The VAS-A consists of a 10 cm horizontal line ranging from 0 to 10, with zero representing the lowest level of anxiety and 10 representing the highest level.
Family Satisfaction in the İntensive Care Unit | 5 minutes
  The scale consists of 24 five-point Likert-type questions and consists of three sub-dimensions: care, decision-making and knowledge. For each statement, respondents mark the most appropriate answer between 1 and 5, ranging from 5 (Excellent) to 1 (Poor). The higher the scores obtained from the scale, the higher the level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided